CLINICAL TRIAL: NCT04254016
Title: Short Term Effects of a Hibiscus Sabdariffa and Stevia Rebaudiana Drink on Cardiac Relaxation and Urinary Albumin Excretion in a Group of Diabetic Type 2 Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Responsible Party: Principal Investigator, CN NGANOU-GNINDJIO, MD, MSc, Dr, Principal investigator, Yaounde Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIBISTEVER
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Benefits of a Hibiscus Sabdariffa and Stevia Rebaudiana Drink in Patients With Type 2 Diabetes Mellitus Before and After 8 Weeks of add-on Therapy
Keywords: Diastolic function; Blood pressure; Diabetes mellitus; Hibiscus Sabdariffa; Stevia Rebaudiana
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-randomized single-arm of HIBISTEVER1 (Experimental): Non-randomized single-arm clinical trial with a before and after design. The study population consisted on all type 2 diabetes mellitus (T2DM) patients with a target population of T2DM patients with HbA1c between 42 to 64mmol/mol (6-8%) with no change in anti-diabetic treatment during the last three months, previous the study.
  The intervention consisted on the administration of Hibiscus-Stevia drink at a dose of 4 mg / kg / day / for Stevia and 4 g / day for Hibiscus for a period of 8 weeks and after meals.
  Interventions: Dietary Supplement: HIBISTEVER1

INTERVENTIONS:
Dietary Supplement: HIBISTEVER1 — During 8 weeks, administration of a Hibiscus-Stevia drink for 8 weeks at a dose of 4 mg / kg / day for Stevia and 4 g / day for Hibiscus. Evaluation will take place the 30th and 60th days.

SUMMARY:
The aim of this study is to evaluate the effects of a Hibiscus Sabdariffa and Stevia Rebaudiana drink on cardiac relaxation and urinary albumin excretion in a group of diabetic type II patients.

DETAILED DESCRIPTION:
The investigators performed a non-randomized single-arm clinical trial with a before and after design, carried out from November 2016 and May 2017.

Intervention consisted of the administration of a Hibiscus-Stevia drink at a dose of 4 mg / kg / day for Stevia and 4 g / day for Hibiscus for a period of 8 weeks. Before and after intervention, the following were done by the participants: bioelectrical impedance analysis (BIA), blood pressure measurements, fasting blood sugar, HbA1c, lipid profiles, liver function tests, kidney function tests, urinary excretion of albumin tests and full blood counts. These were followed by morphological workup including Electrocardiograms (ECGs), transthoracic heart ultrasounds and Ambulatory Blood Pressure Measurements (ABPM), also done before and after intervention.

Clinical evaluation with fasting blood sugar control, blood pressure controls and urinary excretion albumin tests were done at the 30th and 60th days for safety purposes.

ELIGIBILITY:
Inclusion Criteria:

* Known T2DM patients aged above 21years No change in anti-diabetic medication during the last three months HbA1c between 42 to 64mmol/mol (6-8% Clearance of creatinine calculated according to the Modification of Diet in Renal Disease equation> 60ml/min/1.73 m2

Exclusion Criteria:

* Patient already on Hibiscus or stevia supplementation or other herbal medication Drugs that could interact with hibiscus or whose effects may be amplified, as far back as 1 month before study.

Cardiac, renal disease and liver pathologies Sensitivity, intolerance or allergy to hibiscus or stevia Discontinued intervention Withdrawal of consent

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Variation of mitral E' velocity | 8 weeks
  The mitral E' velocity is one of the methods for evaluating diastolic function.

SECONDARY OUTCOMES:
Urinary excretion of albumin | 8 weeks
  Urinary excretion of albumin level
Variation of transmitral flow parameters such as E velocity | 8 weeks
  E (early diastolic filling velocity)
Variation of blood pressure. | 8 weeks
  Change in systolic and diastolic blood pressure by using ABPM (mmHg)
Variation of lipid profile. | 8 weeks
  Change of triglycerides, LDL cholesterol, HDL cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- Yaounde Central Hospital, NAtional Obesity Center, Yaoundé, Cameroon